CLINICAL TRIAL: NCT05440708
Title: REVERT- Liver Cancer: A Phase 1b/2 Multicenter, Open-label Study to Evaluate the Safety and Efficacy of TTI-101 as Monotherapy and in Combination in Participants With Locally Advanced or Metastatic, and Unresectable Hepatocellular Carcinoma
Brief Title: A Study of TTI-101 as Monotherapy and in Combination in Participants With Locally Advanced or Metastatic, and Unresectable Hepatocellular Carcinoma
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Tvardi Therapeutics, Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TVD-101-001H
Record Dates: First submitted 2022-06-27; First posted 2022-07-01 (Actual); Last update posted 2025-10-22 (Actual); Status verified 2025-02

CONDITIONS: Hepatocellular Carcinoma
Keywords: Hepatocellular carcinoma; TTI-101; Pembrolizumab; Atezolizumab; Bevacizumab; revert
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — C188-9 compound; pembrolizumab; atezolizumab; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Cohort A: TTI-101 as a Single Agent (Experimental): Cohort A Phase 1b: Participants will receive various dose levels of TTI-101 as a single agent to determine the RP2D.
  Cohort A Phase 2: Enrollment in Phase 2 may commence with approval from the safety review committee. Participants will be enrolled and treated at the RP2D of TTI-101 as a single agent.
  Interventions: Drug: TTI-101
- Cohort B: TTI-101 in Combination with Pembrolizumab (Experimental): Cohort B Phase 1b: Participants will receive various dose levels of TTI-101 in combination with pembrolizumab to determine the RP2D.
  Cohort B Phase 2: Enrollment in Phase 2 may commence with approval from the safety review committee. Participants will be enrolled and treated at the RP2D of TTI-101 in combination with pembrolizumab.
  Interventions: Drug: TTI-101; Drug: Pembrolizumab
- Cohort C: TTI-101 in Combination with Atezolizumab and Bevacizumab (Experimental): Cohort C Phase 1b: Participants will receive various dose levels of TTI-101 in combination with atezolizumab and bevacizumab to determine the RP2D.
  Cohort C Phase 2: Enrollment in Phase 2 may commence with approval from the safety review committee. Participants will be enrolled and treated at the RP2D of TTI-101 in combination with atezolizumab and bevacizumab.
  Interventions: Drug: TTI-101; Drug: Atezolizumab; Drug: Bevacizumab

INTERVENTIONS:
Drug: TTI-101 — Oral tablet
Drug: Pembrolizumab — Intravenous (IV) infusion
  Other Names: Keytruda®
  Arms: Cohort B: TTI-101 in Combination with Pembrolizumab
Drug: Atezolizumab — Intravenous (IV) infusion
  Other Names: Tecentriq®
  Arms: Cohort C: TTI-101 in Combination with Atezolizumab and Bevacizumab
Drug: Bevacizumab — Intravenous (IV) infusion
  Other Names: Avastin®
  Arms: Cohort C: TTI-101 in Combination with Atezolizumab and Bevacizumab

SUMMARY:
The primary objectives of Cohort A Phase 1b are to evaluate the safety and tolerability of TTI-101 orally administered as a single agent to participants with locally advanced or metastatic, and unresectable Hepatocellular Carcinoma (HCC) and to determine the maximum tolerated dose (MTD) and/or recommended Phase 2 dose (RP2D) of TTI-101 as a single agent.

The primary objectives of Cohort A Phase 2 are to evaluate the safety and tolerability of TTI-101 orally administered as a single agent at the RP2D to participants with locally advanced or metastatic, and unresectable HCC and to assess the preliminary efficacy of TTI-101 as a single agent in participants with locally advanced or metastatic, and unresectable HCC. The secondary objectives of Cohort A Phase 2 are to assess response, progression, survival, and pharmacokinetics.

The primary objectives of Cohorts B and C Phase 1b are to evaluate the safety and tolerability of TTI-101 orally administered in combination with pembrolizumab therapy (Cohort B) and in combination with atezolizumab and bevacizumab therapy (Cohort C) to participants with locally advanced or metastatic, or unresectable HCC and to determine the MTD and/or RP2D of TTI-101 when used in combination with pembrolizumab therapy (Cohort B) and in combination with atezolizumab and bevacizumab therapy (Cohort C).

The primary objectives of Cohorts B and C Phase 2 are to evaluate the safety and tolerability of TTI-101 orally administered in combination with pembrolizumab therapy (Cohort B) and in combination with atezolizumab and bevacizumab therapy (Cohort C) at the RP2D to participants with locally advanced or metastatic, and unresectable HCC and to assess the preliminary efficacy of TTI-101 in combination with pembrolizumab therapy (Cohort B) and in combination with atezolizumab and bevacizumab therapy (Cohort C) to participants with locally advanced or metastatic, and unresectable HCC. The secondary objectives of Cohorts B and C Phase 2 are to assess response, progression, survival, and pharmacokinetics.

ELIGIBILITY:
Inclusion Criteria:

1. Able to understand and willing to provide informed consent and able to comply with the study procedures and restrictions.
2. Age ≥18 years at the time of informed consent.
3. Have histologically or radiographically (Liver Imaging Reporting and Data Systems category 5) confirmed diagnosis of locally advanced or metastatic, and unresectable HCC. Participants without cirrhosis require histological confirmation.
4. Cohorts A and B only: Willing to provide a representative fresh tumor tissue specimen prior to enrollment. The fresh tumor specimen must be obtained after progression on the prior therapy. No biopsy is required for participants in Cohort C.
5. Measurable disease as per RECIST Version 1.1. Participants who received prior local therapy are eligible provided the target lesion(s) have not been previously treated with local therapy or the target lesion(s) within the field of local therapy have subsequently progressed in accordance with RECIST Version 1.1.
6. Able to swallow tablets.
7. Has an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
8. Has adequate hematologic and organ function as defined by the following local laboratory values at screening:

   * Absolute neutrophil count (ANC) ≥1.5 × 10^9/L (1500/μL) without granulocyte colony-stimulating factor support.
   * Lymphocyte count ≥0.5 × 10^9/L (500/μL).
   * Platelet count ≥75 × 10^9/L (75,000/μL) without transfusion.
   * Hemoglobin ≥90 g/L (9 g/dL). Participants may be transfused to meet this criterion.
   * Serum albumin ≥28 g/L (2.8 g/dL).
   * AST, ALT, and alkaline phosphatase (ALP) ≤5 × upper limit of normal (ULN).
   * Serum bilirubin ≤2 mg/dL.
   * Adequate renal function defined as either:

     * creatinine clearance ≥40 mL/min calculated using the Cockcroft-Gault formula, or
     * 24-hour urine collection.
9. Prothrombin time/international normalized ratio (PT/INR) and activated partial thromboplastin time (aPTT) ≤2 × ULN, except for participants receiving anticoagulation therapy.
10. Child-Pugh class A or B7 within 7 days prior to enrollment.
11. Females of childbearing potential (ie, ovulating, premenopausal, and not surgically sterile) must:

    * Have a negative serum pregnancy test at screening.
    * Not be breastfeeding or lactating.
    * Agree to use a highly effective method of birth control for the duration of the study and for at least 30 days after the last dose in the study. Effective forms of birth control include barrier methods used in conjunction with a spermicidal agent (according to standard local practices), nonhormonal intrauterine devices, or permanent sterilization.
12. Males must:

    * Agree to use a condom for at least 30 days after the last dose in the study even if vasectomized in order to prevent delivery of the drug via seminal fluid.
    * Agree to abstain from sperm donation through 30 days after administration of the last dose of the study treatment.
    * Unless surgically sterile, males with female partners of childbearing potential must agree to use 2 methods of acceptable birth control for at least 30 days after the last dose in the study. Effective forms of birth control include barrier methods used in conjunction with a spermicidal agent (according to standard local practices), nonhormonal intrauterine devices in female partners, or permanent sterilization.

    Cohort A:
13. In addition to the general inclusion criteria, participants enrolled in Cohort A must have demonstrated objective progression on up to 3 prior lines of systemic antitumor drug therapy.

    Cohort B:
14. In addition to the general inclusion criteria, participants enrolled in Cohort B must have demonstrated objective progression following at least 2 cycles of first-line anti-PD-1 or anti-PD-L1 monotherapy or combination therapy. Participants may have received no more than one line of prior systemic therapy.
15. Agree to use contraception as specified in the general inclusion criteria for at least 4 months following the last dose of pembrolizumab in accordance with the approved prescribing information.

    Cohort C:
16. In addition to the general inclusion criteria, participants enrolled in Cohort C must be naïve to systemic treatment for locally advanced or metastatic, and unresectable HCC.
17. Must have had an evaluation (gastroduodenoscopy) for the presence of varices within 6 months prior to initiation of bevacizumab therapy.
18. Agree to use contraception as specified in the general inclusion criteria for at least 5 months after the last dose of atezolizumab and at least 6 months after the last dose of bevacizumab in accordance with the approved prescribing information.

Exclusion Criteria:

1. Pregnant or breastfeeding.
2. Known fibrolamellar HCC, sarcomatoid HCC, or mixed cholangiocarcinoma and HCC.
3. History of leptomeningeal disease.
4. Previous treatment of the current malignancy with a signal transducer and activator of transcription (STAT) inhibitor.
5. Previous therapy with:

   1. Standard therapy including chemotherapy, immunotherapy, biologic therapy, or any other anticancer therapy within 28 days (or 5 elimination half-lives for non-cytotoxics, whichever is shorter) of Cycle 1 Day 1 (6 weeks for nitrosoureas or mitomycin).
   2. Any investigational agent within 28 days (or 5 elimination half-lives for a non-cytotoxic investigational therapy, whichever is shorter) of Cycle 1 Day 1 or 5 half-lives for a small molecule/targeted therapy.
6. Extensive prior radiotherapy to more than 30% of bone marrow reserves, or prior bone marrow/stem cell transplantation within 5 years from enrollment.
7. Herbal preparations are not allowed throughout the study. These herbal medications include but are not limited to St. John's wort, kava, ephedra (mahung), gingko biloba, dehydroepiandrosterone (DHEA), yohimbe, saw palmetto, and ginseng. Participants should stop using herbal medications 7 days prior to the first dose of study treatment.
8. Is not fully recovered from all coronavirus disease 2019 (COVID-19)-related symptoms for 2 weeks prior to Cycle 1 Day 1, if previously tested positive for COVID-19.
9. Ongoing toxicity (except alopecia) due to a prior therapy, unless returned to baseline or Grade 1 or less.
10. Has had major surgery within 3 weeks prior to starting investigational product (IP) or has not recovered from major side effects due to surgery.
11. Significantly impaired cardiac function such as unstable angina pectoris, congestive heart failure with New York Heart Association Class III or IV, myocardial infarction within the last 12 months prior to study entry; serious arrhythmia (including QTc prolongation of >450 ms for males and >470 ms for females and/or pacemaker) or prior diagnosis of congenital long QT syndrome or left ventricular ejection fraction <50% on screening echocardiogram.
12. Pleural effusion, pericardial effusion, or ascites requiring recurrent drainage procedures (once monthly or more frequently). Participants with indwelling catheters for control of effusions or ascites are allowed.
13. History of cerebrovascular accident or stroke within the previous 2 years.
14. History of hepatic encephalopathy.
15. Uncontrolled or symptomatic hypercalcemia (ionized calcium >1.5 mmol/L, calcium >12 mg/dL, or corrected serum calcium >ULN).
16. Evidence of bleeding diathesis or significant coagulopathy (in the absence of therapeutic anticoagulation).
17. History of Grade 3 or 4 allergic reactions attributed to compounds of similar chemical or biologic composition as TTI-101 (hydroxyl-naphthalene sulfonamides).
18. Known active metastases in the central nervous system (unless stable by brain imaging studies for at least 1 month without evidence of cerebral edema and no requirements for corticosteroids or anticonvulsants).
19. History of difficulty swallowing oral medications, malabsorption, or other chronic gastrointestinal disease or conditions that may hamper compliance and/or absorption of the IP.
20. Has a known history of human immunodeficiency virus (HIV) infection.
21. Participants with chronic hepatitis B virus (HBV) infection, unless screening viral load <500 IU/mL on stable doses of antiviral therapy. Note: Participants with chronic hepatitis C virus (HCV) infection are allowed to enroll into the study but do not have a defined maximum viral load requirement for study entry. Participants with both HBV and HCV infection are excluded unless they have negative HCV ribonucleic acid (RNA).
22. History of malignancy other than HCC within 3 years prior to screening, with the exception of malignancies with a negligible risk of metastasis or death (eg, 5-year overall survival [OS] rate >90%), such as adequately treated carcinoma in situ of the cervix, non-melanoma skin carcinoma, localized prostate cancer, ductal carcinoma in situ, or Stage I uterine cancer.
23. Has any other concurrent severe and/or uncontrolled medical condition that would, in the investigator's judgment, cause unacceptable safety risks, contraindicate participation in the clinical study, or compromise compliance with the protocol such as:

    * Chronic pancreatitis.
    * Active untreated or uncontrolled fungal, bacterial, or viral infections (including COVID-19), sepsis, etc.
    * Acute and chronic, active infectious disorders including viral and nonmalignant medical illnesses that are uncontrolled or whose control may be jeopardized by the complications of this study therapy.
24. Is unable to understand and to comply with study instructions and requirements.

    Cohort B:

    In addition to the general exclusion criteria, participants enrolled in Cohort B must fulfill the following additional exclusion criteria:
25. Discontinued prior treatment with anti-PD-1 or anti-PD-L1 for any reason other than disease progression.

    Cohort C:

    In addition to the general exclusion criteria and Cohort B criteria, participants enrolled in Cohort C must fulfill the following additional exclusion criteria:
26. Inadequately controlled arterial hypertension (defined as systolic blood pressure [BP] ≥150 mmHg and/or diastolic BP ≥100 mmHg), based on an average of ≥3 BP readings on ≥2 sessions.
27. Participant has received prior systemic chemotherapy for locally advanced or metastatic and/or unresectable HCC. However, participant may have received either neo-adjuvant or adjuvant chemotherapy as long as it was completed at least 6 months prior to the first dose of study treatment.
28. Untreated or incompletely treated esophageal and/or gastric varices with bleeding or high risk for bleeding and a prior bleeding event due to esophageal and/or gastric varices within 6 months prior to initiation of study treatment.
29. Urine dipstick for proteinuria ≥2+ at screening. If a 24-hour urine collection shows <1 g of protein in 24 hours, the participant is eligible.
30. Current or recent (within 10 days of first dose of study treatment) use of aspirin (>325 mg/day) or treatment with dipyridamole, ticlopidine, clopidogrel, and cilostazol.
31. Current or recent (within 10 days prior to study treatment start) use of full-dose oral or parenteral anticoagulants. Prophylactic anticoagulants (eg, low-dose warfarin with target INR <1.5 × ULN or low-dose low molecular weight heparin) are allowed.
32. Core biopsy or other minor surgical procedure, excluding placement of a vascular access device, within 3 days prior to the first dose of bevacizumab.
33. History of gastrointestinal perforation or evidence of abdominal free air not explained by paracentesis or recent surgical procedure.
34. Metastatic disease that involves major airways or blood vessels. Participants with portal or hepatic vein involvement are not excluded.
35. Participant has experienced any of the following within 6 months prior to enrollment: arterial thromboembolic event (including myocardial infarction, coronary arterial disease, transient ischemic attack, stroke, etc), congestive heart failure, hemoptysis, or pulmonary embolism.
36. Participant has experienced a fistula.

    Cohorts B and C:

    In addition to the general exclusion criteria and the cohort-specific criteria listed above, participants enrolled in Cohorts B and C must fulfill the following additional exclusion criteria:
37. Treatment with a live, attenuated vaccine within 4 weeks prior to initiation of study treatment, or anticipation of need for such a vaccine during pembrolizumab treatment or within 5 months after the last dose of pembrolizumab treatment.
38. Active or history of immune-mediated disease or immune deficiency, including, but not limited to, myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, antiphospholipid antibody syndrome, Wegener granulomatosis, Sjögren's syndrome, Guillain-Barré syndrome, or multiple sclerosis, with the following exceptions:

    * Participants with a history of autoimmune-related hypothyroidism who are on thyroid-replacement hormone are eligible for the study.
    * Participants with controlled Type 1 diabetes mellitus who are on an insulin regimen are eligible for the study.
    * Participants with eczema, psoriasis, lichen simplex chronicus, or vitiligo with dermatologic manifestations only (eg, participants with psoriatic arthritis are excluded) are eligible for the study provided all of the following conditions are met:

      * Rash must cover <10% of body surface area.
      * Disease is well controlled at baseline and requires only low-potency topical corticosteroids.
      * No occurrence of acute exacerbations of the underlying condition requiring psoralen plus ultraviolet A radiation, methotrexate, retinoids, biologic agents, oral calcineurin inhibitors, or high-potency or oral corticosteroids within the previous 12 months.
39. History of idiopathic pulmonary fibrosis, organizing pneumonia (eg, bronchiolitis obliterans), drug-induced pneumonitis, or idiopathic pneumonitis, or evidence of active pneumonitis on screening chest computed tomography (CT) scan. History of radiation pneumonitis in the radiation field (fibrosis) is permitted.
40. Treatment with systemic immunosuppressive medication (including, but not limited to, corticosteroids, cyclophosphamide, azathioprine, methotrexate, thalidomide, and anti-tumor necrosis factor α [TNF-α] agents) within 2 weeks prior to initiation of study treatment. Participants receiving low-dose corticosteroids (equivalent of prednisone 10 mg/day or lower) or who receive pulse corticosteroids due to intravenous (IV) contrast allergy are not excluded.
41. Active tuberculosis.
42. Severe infection within 4 weeks prior to initiation of study treatment, including, but not limited to, hospitalization for complications of infection, bacteremia, or severe pneumonia.
43. Treatment with therapeutic oral or IV antibiotics within 2 weeks prior to initiation of study treatment. Participants receiving prophylactic antibiotics (eg, to prevent a urinary tract infection or chronic obstructive pulmonary disease exacerbation) are eligible for the study.
44. Prior allogeneic stem cell or solid organ transplantation.
45. History of severe allergic anaphylactic reactions to chimeric or humanized antibodies or fusion proteins.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 178 (Estimated)
Dates: Start 2023-03-23 (Actual); Primary Completion 2026-06-29 (Estimated); Study Completion 2027-06-28 (Estimated)

PRIMARY OUTCOMES:
Incidence of Adverse Events (AE) | Up to approximately 20 months
  An AE is any untoward medical occurrence in a participant or clinical study participant administered a pharmaceutical product and which does not necessarily have a causal relationship with this treatment. Any clinically significant changes between baseline and postbaseline laboratory assessments, electrocardiograms (ECGs), vital signs and physical examinations will be recorded as AEs.
Incidence of Serious Adverse Events (SAE) | Up to approximately 18 months
Phase 2: Overall Response Rate (ORR) to TTI-101 | Up to approximately 18 months
  ORR (calculated as Partial Response [PR] + Complete Response [CR]) using RECIST Version 1.1.

SECONDARY OUTCOMES:
Phase 1b: Overall Response Rate (ORR) to TTI-101 | Up to approximately 18 months
  Defined as complete response (CR) + partial response (PR) measured in all participants using RECIST Version 1.1.
Duration of Response (DoR) to TTI-101 | Up to approximately 18 months
Disease Control Rate (DCR) to TTI-101 | Up to approximately 18 months
Duration of Disease Control (DDC) to TTI-101 | Up to approximately 18 months
Time to Tumor Progression (TTP) to TTI-101 | Up to approximately 18 months
Best Overall Response (BOR) to TTI-101 | Up to approximately 18 months
Progression Free Survival (PFS) to TTI-101 at 6 months | Month 6
Progression Free Survival (PFS) to TTI-101 at 12 months | Month 12
Maximum Observed Plasma Concentration (Cmax) of TTI-101 | Cycle 2 Day 15 (cycle is 21 days)
Time of Maximum Observed Plasma Concentration (Tmax) of TTI-101 | Cycle 2 Day 15 (cycle is 21 days)
Area Under the Plasma Concentration-Time Curve from Time 0 to Time t (AUC0-t) of TTI-101 | Cycle 2 Day 15 (cycle is 21 days)
Terminal Elimination Half-life (t1/2) of TTI-101 | Cycle 2 Day 15 (cycle is 21 days)
Area Under the Plasma Concentration-time Curve from Time 0 to Infinity (AUC0-∞) of TTI-101 | Cycle 2 Day 15 (cycle is 21 days)
Apparent Plasma Clearance (CL/F) of TTI-101 | Cycle 2 Day 15 (cycle is 21 days)
Cohort A and Cohort B: Pharmacodynamics of TTI-101 as Measured By Change from Baseline in Percentage of Phosphorylated Signal Transducer and Activator of Transcription 1 (pY-STAT1) Positive Cells in Tumor Biopsy Samples | Baseline up to approximately 18 months
Cohort A and Cohort B: Pharmacodynamics of TTI-101 as Measured By Change from Baseline in Percentage of Phosphorylated Signal Transducer and Activator of Transcription 3 (pY-STAT3) Positive Cells in Tumor Biopsy Samples | Baseline up to approximately 18 months
Cohort A and Cohort B: Pharmacodynamics of TTI-101 as Measured By Change from Baseline in Percentage of Phosphorylated Signal Transducer and Activator of Transcription 5 (pY-STAT5) Positive Cells in Tumor Biopsy Samples | Baseline up to approximately 18 months

CONTACTS AND LOCATIONS:
Locations (21):
- United States (21):
  - The Kirklin Clinic of University of Alabama Birmingham Hospital, Birmingham, Alabama
  - University of California San Diego, La Jolla, California
  - Norris Comprehensive Cancer Center, Los Angeles, California
  - University of California Irvine Medical Center, Orange, California
  - University of Colorado Hospital - Anschutz Medical Campus, Aurora, Colorado
  - Georgetown Lombardi Comprehensive Cancer Center, Washington D.C., District of Columbia
  - Moffitt Cancer Center, Tampa, Florida
  - The Sidney Kimmel Comprehensive Cancer Center, Baltimore, Maryland
  - University of Michigan Rogel Cancer Center, Ann Arbor, Michigan
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Washington University in St. Louis, St Louis, Missouri
  - Memorial Sloan Kettering Cancer Center - New York, New York, New York
  - Cleveland Clinic Lerner College of Medicine, Cleveland, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Harold C. Simmons Comprehensive Cancer Center, Dallas, Texas
  - DHR Health Institute for Research & Development, Edinburg, Texas
  - University of Texas MD Anderson Cancer Center, Houston, Texas
  - University of Texas Health Science Center - San Antonio, San Antonio, Texas
  - Virginia Mason Medical Center, Seattle, Washington
  - Summit Cancer Centers - North Spokane, Spokane, Washington
  - Froedtert and Medical College of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No